CLINICAL TRIAL: NCT05982717
Title: Epidemiology of Dravet and Lennox-Gastaut Syndromes in Spain
Brief Title: A Study to Gather Information About Overall Occurrence and New Cases of Dravet and Lennox-Gastaut Syndromes in Children, Teenagers and Adults in Spain
Acronym: DRALEGA
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-935-5003
Record Dates: First submitted 2023-07-28; First posted 2023-08-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Dravet Syndrome (DS); Lennox-Gastaut Syndrome (LGS)
Keywords: Drug Therapy
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With DS or LGS: Participants with a medical record of diagnosis with either DS or LGS that are treated in the participating hospitals and reside in the reference area of these hospitals will be included and data will be retrospectively collected for the period between 01 January 2021 to 31 December 2022.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
The main aims of this study are to gather information about how many children, teenagers and adults in Spain have been diagnosed with Dravet syndrome and Lennox-Gastaut syndrome as well as to learn about the number of new Dravet syndrome and Lennox-Gastaut syndrome cases in persons in Spain.

Participants' data will be taken from their medical records (charts), which were already collected as a part of their routine care in public hospitals in Spain between 01 January 2021 and 31 December 2022.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective study of participants from Spain with DS and LGS at public hospitals. The participants will be identified from their medical charts or hospital records and those who meet the eligibility criteria will be included.

This multi-center trial will be conducted in Spain. Data will be retrospectively collected for the observation period between 01 January 2021 to 31 December 2022. The total duration of the study is approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

A. Diagnosis criteria for DS:

• All the following criteria must be met: i. Seizures onset within 1-20 months (usually within the first year of life). ii. Normal initial development prior to presentation (no cognitive or behavioural disability before the onset of seizures) followed by behaviour and cognitive impairment.

iii. Recurrent focal clonic (hemiclonic) febrile and afebrile seizures (which often alternate sides from seizure to seizure), focal to bilateral tonicclonic, and/or generalized clonic seizures.

• And at least one of the following criteria must be met: i. Emergence of other seizure type, including atypical absence seizures, myoclonic seizures, atonic seizures, or non-tonic-clonic status epilepticus between 1-4 years.

ii. Seizures triggered by fever due to illness or vaccinations, hot baths, sudden temperature changes, high level of activity, or by strong lighting or exposure to certain visual patterns.

iii. Mutations or copy number variants in the SCN1A gene.

B. Diagnosis criteria for LGS:

Given the uncertainties associated with the diagnosis of this condition, two different criteria will be used, a stricter criterion, intended to identify "pure" Lennox-Gastaut syndrome participants, and a wider criterion, intended to also include the so-called Lennox-Gastaut-like participants.

Lennox-Gastaut syndrome - stricter criteria:

• All the following criteria must be met: i. Seizures onset before 18 years of age, typically from 1 to 8 years. ii. Progressive development/cognition impairment after seizures onset. iii. Tonic seizures. iv. At least one additional seizure: generalised tonic-clonic seiures, atypical absence seizures, atonic seizures, myoclonic seizures, focal impaired awareness, epileptic spams, or non-convulsive status epilepticus v. Slow (<2.5 hertz [Hz]) spike-and-wave EEG pattern. vi. Paroxysmal fast activity (10 Hz or greater) in sleep.

Lennox-Gastaut syndrome - wider criteria:

* At least one the following criteria must be met:

  i. Tonic seizures. ii. Multiple types of seizures, including generalised tonic-clonic seizures, atypical absence seizures, atonic seizures, myoclonic seizures, myoclonic-atonic seizures, focal seizures, epileptic spams, or nonconvulsive status epilepticus.
* And at least one the following criteria must be met:

  i. Slow (<2.5 Hz) spike-and-wave EEG pattern. ii. Paroxysmal fast activity (10 Hz or greater) in sleep.
* And at least two of the following criteria must be met:

  i. Seizures onset before 18 years of age, typically from 1 to 8 years. ii. Progressive development/cognition impairment after seizures onset. iii. Development/cognition impairment starts prior to seizures onset. iv. History of Infantile epileptic spasms syndrome (IESS), West or Ohtahara syndromes.

Exclusion Criteria

1. Participants with epileptic condition other than DS or LGS.
2. Participants with DS or LGS not residents in the reference area of the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with DS or LGS at public hospitals in Spain will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
One-Year Period Prevalence of DS | Up to 12 months
  Number of participants with DS over a period of one year will be assessed.
Incidence of DS | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Number of new participants diagnosed annually with DS yearly.
One-Year Period Prevalence of LGS Based on Stricter Diagnosis Criterion | Up to 12 months
  Number of participants with LGS over a period of one year based on stricter diagnosis criterion will be assessed.
Incidence of LGS Based on Stricter Diagnosis Criterion | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Number of new participants diagnosed annually with LGS based on stricter diagnosis criterion.

SECONDARY OUTCOMES:
One-Year Period Prevalence of LGS Based on Wider Diagnosis Criterion | Up to 12 months
  Number of participants with LGS over a period of one year based on wider diagnosis criterion will be assessed.
Incidence of LGS Based on Wider Diagnosis Criterion | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Number of new participants diagnosed annually with LGS based on wider diagnosis criterion.
One-Year Period Prevalence of Paediatric DS | Up to 12 months
  Number of participants with paediatric DS over a period of one year will be assessed.
One-Year Period Prevalence of Paediatric LGS Based on Stricter and Wider Diagnoses Criteria | Up to 12 months
  Number of participants with paediatric LGS over a period of one year based on stricter and wider diagnoses criteria will be assessed.
One-Year Period Prevalence of Adult DS | Up to 12 months
  Number of participants with adult DS over a period of one year will be assessed.
One-Year Period Prevalence of Adult LGS Based on Stricter and Wider Diagnoses Criteria | Up to 12 months
  Number of participants with adult LGS over period of one year based on stricter and wider diagnoses criteria will be assessed.
Incidence of Paediatric DS | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Number of new paediatric participants diagnosed annually with DS.
Incidence of Paediatric LGS Based on Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Number of new paediatric participants diagnosed annually with LGS based on stricter and wider diagnoses criteria.
Incidence of Adult DS | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Number of new adult participants diagnosed annually with DS.
Incidence of Adult LGS Based on Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Number of new adult participants diagnosed annually with LGS based on stricter and wider diagnoses criteria.
DS Categorized Based on Gender Distribution | Up to 12 months
LGS Categorized Based on Gender Distribution According to Stricter and Wider Diagnoses Criteria | Up to 12 months
DS Categorized Based on Age Distribution | Up to 12 months
LGS Categorized Based on Age Distribution According to Stricter and Wider Diagnoses Criteria | Up to 12 months
DS Categorized Based on Gender Distribution at Diagnosis | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Annually diagnosed DS participants will be categorized based on gender distribution at diagnosis.
LGS Categorized Based on Gender Distribution at Diagnosis According to Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Annually diagnosed LGS participants will be categorized based on gender distribution at diagnosis.
DS Categorized Based on Age Distribution at Diagnosis | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Annually diagnosed DS participants will be categorized based on age distribution at diagnosis.
LGS Categorized Based on Age Distribution at Diagnosis According to Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Annually diagnosed LGS participants will be categorized based on age distribution at diagnosis.
DS Categorized Based on Gender Distribution at Symptoms Onset | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Annually diagnosed DS participants will be categorized based on gender distribution at symptoms onset.
LGS Categorized Based on Gender Distribution at Symptoms Onset According to Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Annually diagnosed LGS participants will be categorized based on gender distribution at symptoms onset.
DS Categorized Based on Age Distribution at Symptoms Onset | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Annually diagnosed DS participants will be categorized based on age distribution at symptoms onset.
LGS Categorized Based on Age Distribution at Symptoms Onset According to Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Annually diagnosed LGS participants will be categorized based on age distribution at symptoms onset.
Diagnosis Delay for Participants With DS | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Diagnosis delay is defined as time from symptoms onset to diagnosis.
Diagnosis Delay for Participants With LGS Based on Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)
  Diagnosis delay is defined as time from tonic seizures onset to electroencephalography (EEG) confirmation.
Participants With DS: Ratio of Participants Genetically (Sodium Channel Protein Type 1 Subunit Alpha [SCN1A] Mutation) and Clinically Diagnosed Versus Participants Clinically Diagnosed Only | At two different 12 month periods (in consecutive years at Months 12 and 24)
Participants With LGS: Number of Participants Distributed According to Aetiologies Based on Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)
Participants With DS: Number of Participants With Different Types of Comorbidities at Diagnosis | At two different 12 month periods (in consecutive years at Months 12 and 24)
Participants With LGS: Number of Participants With Different Types of Comorbidities at Diagnosis Based on Stricter and Wider Diagnoses Criteria | At two different 12 month periods (in consecutive years at Months 12 and 24)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- Spain (4):
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - H. Universitario Infantil Niño Jesús, Madrid
  - H. Universitario La Paz, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/b7d67115dd3848ae?idFilter=%5B%22TAK-935-5003%22%5D